CLINICAL TRIAL: NCT03941366
Title: Treatment of T2-T3/NO-N+ Adenocarcinoma of the Rectum by Neoadjuvant Chemotherapy (FOLFOX) Followed by Preoperative Chemo (5FU/Capecitabine)-Radio Therapy (CRT) With Transanal Local Excision for Complete Responders
Brief Title: Treatment of Adenocarcinoma of the Rectum With Transanal Local Excision for Complete Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Amr Aref, Director, Radiation Oncology, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 866142
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients in the trial receive the intervention and are followed prospectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Chemotherapy and Follow-up Surgery (Other): All patients will receive standard of care therapy and based upon their response will either receive transanal local resection or full resection, based on pathologic response.
  Interventions: Procedure: Standard of care chemotherapy with the change for avoidance of extensive surgery

INTERVENTIONS:
Procedure: Standard of care chemotherapy with the change for avoidance of extensive surgery — All treatments (chemotherapy, radiation, surgery) are standard of care; however, the timing of the procedures is altered to allow for the possibility of local excision instead of more extensive surgery.

SUMMARY:
The current standard of care for rectal cancer has diminished local recurrence and enhanced survival. Quality of life, however, remains poor for many patients and the probability of distant recurrence is high. In this study, we will attempt to reduce the distant recurrence rate and improve quality of life by making changes in the timing and administration of chemotherapy and radiation and doing less invasive rectal surgery when indicated.

DETAILED DESCRIPTION:
The purpose of the study is to determine if neo-adjuvant FOLFOX therapy and lengthening the time interval between neo-adjuvant chemotherapy and transanal local excision will increase the percentage of patients with pathologic complete remission.

This is a prospective pilot study to examine the impact of two variables: 1) addition of neo-adjuvant FOLFOX chemotherapy, and 2) increasing the time interval between completion of chemo-radiotherapy and subsequent surgery, on the rate of achieving pathologic complete remission with avoidance of radical resection while maintaining an excellent local control with improvement of quality of life.

All procedures in this study are standard of care, the study question relates to the use of neo-adjuvant FOLFOX and the timing between the end of radiation and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of rectal invasive adenocarcinoma
3. Tumor in the low or mid rectum (up to 11 cm from the anal verge)
4. Clinical stage T3/N0-N1M0. Patients with low T2 who will need abdominal perineal resection are also eligible.

1. Clinical staging will be estimated based on the combination of the following assessments:

1. Physical examination by the primary surgeon
2. Computed Tomography or Positron Emission Tomography/Computed Tomography scan of chest, abdomen and pelvis
3. Pelvic MRI and endoscopic ultrasound

Exclusion Criteria:

* Less than 18 years of age
* Do not complete informed consent
* Pregnant women

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-02-26 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 18 months
  Percent of patients who achieve complete remission
Partial remission | 18 months
  Percent of patients who achieve partial remission
Disease progression | 18 months
  Percent of patients with disease progression
Local resection | 18 months
  Percent of patients who require local resection only

SECONDARY OUTCOMES:
Patient quality of life | 18 months
  Quality of life score on questionnaire
Patient health status | 18 months
  Patient self-reported health status

CONTACTS AND LOCATIONS:
Overall Officials: Amr Aref, MD, Principal Investigator — Ascension SME
Locations (1):
- Ascension St. John Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No